CLINICAL TRIAL: NCT00260975
Title: A Prospective, Longitudinal Investigation of the Neuropsychological and Psychosocial Effects of Cancer Therapy
Brief Title: Study of the Effects of Chemotherapy on Memory and Other Mental Functions in Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1999232-01H
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; hormonal therapy; cognitive function; chemo fog
MeSH Terms: conditions — Breast Neoplasms; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chemotherapy patients: Breast cancer patients treated with adjuvant chemotherapy of various types.
- Hormonal patients: Breast cancer patients treated with adjuvant hormonal therapy but not chemotherapy.

SUMMARY:
Many breast cancer patients treated with chemotherapy complain of problems with concentration and memory. This has been referred to as chemo fog. The current study is investigating this phenomenon by measuring mental function of breast cancer patients prior to and after exposure to chemotherapy, and by comparing mental function in those patients who receive chemotherapy and those who do not.

DETAILED DESCRIPTION:
Many breast cancer patients treated with chemotherapy complain of problems with concentration and memory. This has been referred to as chemo fog. The current study will investigate this phenomenon by measuring neuropsychological functioning in early stage breast cancer patients prior to and after exposure to chemotherapy, and by comparing change in cognitive function in patients who receive chemotherapy to similar breast cancer patients receiving hormonal therapy only.

ELIGIBILITY:
Inclusion Criteria:

* stage I or II breast cancer; woman; 50-65 years old; post-menopausal

Exclusion Criteria:

* history of previous cancer or chemotherapy; significant neurological or psychiatric history

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2001-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Collins, Principal Investigator — OHRI

REFERENCES:
- [Result] Stewart A, Collins B, Mackenzie J, Tomiak E, Verma S, Bielajew C. The cognitive effects of adjuvant chemotherapy in early stage breast cancer: a prospective study. Psychooncology. 2008 Feb;17(2):122-30. doi: 10.1002/pon.1210. PMID 17518411
- [Result] Collins B, Mackenzie J, Stewart A, Bielajew C, Verma S. Cognitive effects of chemotherapy in post-menopausal breast cancer patients 1 year after treatment. Psychooncology. 2009 Feb;18(2):134-43. doi: 10.1002/pon.1379. PMID 18551510
- [Result] Collins B, Mackenzie J, Stewart A, Bielajew C, Verma S. Cognitive effects of hormonal therapy in early stage breast cancer patients: a prospective study. Psychooncology. 2009 Aug;18(8):811-21. doi: 10.1002/pon.1453. PMID 19085975